CLINICAL TRIAL: NCT05923190
Title: A Pilot Trial of Enfortumab Vedotin Schedule De-escalation in Metastatic Urothelial Carcinoma
Brief Title: Enfortumab Vedotin Schedule De-escalation in Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1008; GU-217 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enfortumab vedotin (EV) monotherapy (Active Comparator): EV will be administered at standard dose of 1.25 mg/kg IV on days 1, 8 and 15 of a 28-day cycle for 3 cycles.
  First schedule de-escalation of EV will occur in patients with disease control per RECIST v1.1 (complete response/partial response/stable disease) on their first scan in the EV at 12 weeks. In these patients, EV will be administered on days 1 and 15 of a 28-day cycle.
  Second schedule de-escalation of EV will occur in patients with disease control per RECIST v1.1 (complete response/partial response/stable disease) on their second scan in the EV monotherapy (at 24 weeks). EV will be administered on day 1 of a 21-day cycle.
  Interventions: Drug: Enfortumab vedotin
- EV/pembrolizumab (Experimental): EV will be administered at standard dose of 1.25 mg/kg IV on days 1 and 8 with pembrolizumab 200 mg IV on day 1 of a 21-day cycle for 6 cycles. Radiographic assessment will be conducted every 9 weeks.
  Schedule de-escalation of EV will occur in patients with disease control per RECIST v1.1 (complete response/partial response/stable disease) on their first scan in the EV/pembrolizumab arm at 9 weeks. In these patients EV and pembrolizumab will be administered on day 1 of a 21-day cycle.
  Interventions: Drug: Enfortumab vedotin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Enfortumab vedotin — EV will be administered at standard dose of 1.25 mg/kg IV on days 1 and 8 with pembrolizumab 200 mg IV on day 1 of a 21-day cycle for 6 cycles
Drug: Pembrolizumab — Pembrolizumab will be administered on day 1 of a 21-day cycle
  Arms: EV/pembrolizumab

SUMMARY:
This is a non-randomized two arm open-label phase 2 pilot study in adult subjects with locally advanced or metastatic urothelial cancer. The study will investigate an alternative administration schedule of EV given as monotherapy and in combination with pembrolizumab.

DETAILED DESCRIPTION:
This is a non-randomized two arm open-label phase 2 pilot study in adult subjects with locally advanced or metastatic urothelial cancer. The study will investigate an alternative administration schedule of EV given as monotherapy and in combination with pembrolizumab. Approximately 50 patients will be enrolled to the main EV monotherapy cohort who are scheduled to receive EV as standard of care. Additionally, an exploratory arm will enroll 20 patients with metastatic urothelial cancer who are scheduled to receive EV in combination with pembrolizumab as standard of care. All subjects will have histologically and radiographically confirmed locally advanced or metastatic urothelial carcinoma, Eastern Cooperative Oncology Group (ECOG) performance status 0-2, and meet baseline laboratory data as outlined in the section 4.1.

ELIGIBILITY:
Inclusion Criteria:

EV monotherapy main cohort:

* Patients must have histologically and radiographically confirmed locally advanced or metastatic urothelial carcinoma.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v1.1
* Planned to receive EV as standard treatment for advanced urothelial cancer
* ECOG performance status 0-2
* Prior systemic therapy must have completed at least 14 days prior to initiating therapy.
* Age > 18 years.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Archival tumor biospecimen (when available) must be procured for correlative evaluation. If tumor tissue is not available or accessible despite good faith efforts, patient may still be treated on study. Formalin-fixed paraffin-embedded [FFPE] tissue block(s) or at least 15 unbaked, unstained slides are required. Tissue samples taken from a metastatic lesion prior to the start of screening are acceptable.
* Normal organ and marrow function as defined below.

  * Absolute neutrophil count > 1,000/mm3 unless patient has constitutional neutropenia
  * Platelets > 100,000/ul
  * Hemoglobin > 8.0 g/dL
  * Alanine transaminase (ALT) and aspartate transaminase (AST) <2.5X upper limit of normal (ULN) or <3.5X ULN if liver metastases
  * Creatinine Clearance >20 ml/min

EV/pembrolizumab arm:

* Patients must have histologically and radiographically confirmed locally advanced or metastatic urothelial carcinoma.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v1.1
* Planned to receive EV/pembrolizumab as standard treatment for advanced urothelial cancer
* ECOG performance status 0-2
* Prior systemic therapy must have completed at least 14 days prior to initiating therapy.
* Age > 18 years.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Archival tumor biospecimen (when available) must be procured for correlative evaluation. If tumor tissue is not available or accessible despite good faith efforts, patient may still be treated on study. Formalin fixed, paraffin embedded [FFPE] tissue block(s) or at least 15 unbaked, unstained slides are required. Tissue samples taken from a metastatic lesion prior to the start of screening are acceptable.
* Normal organ and marrow function as defined below.

  * Absolute neutrophil count > 1,000/mm3 unless patient has constitutional neutropenia
  * Platelets > 100,000/ul
  * Hemoglobin > 8.0 g/dL
  * ALT and AST <2.5X ULN or <3.5X ULN if liver metastases
  * Creatinine Clearance >20 ml/min

Exclusion Criteria:

Both EV monotherapy and EV/pembrolizumab arms:

* Patients who have received prior monomethyl auristatin E (MMAE)-based antibody-drug conjugates (ADCs) for urothelial cancer.
* Grade 2 or higher baseline sensory or motor neuropathy.
* Uncontrolled diabetes (HbA1c >8%)
* Patients with uncontrolled and untreated central nervous system (CNS) metastases.

  * Prior radiation to CNS metastases is permitted.
  * Prior history of CNS disease that has responded to previous systemic therapy is permitted only if no recurrence.
  * Patient should not have leptomeningeal disease
  * CNS metastases have been clinically stable for at least 6 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis.
  * If requiring steroid treatment for CNS metastases, the patient is on stable dose < 20 mg/day of prednisone or equivalent for at least 2 weeks prior to starting treatment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active untreated infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with a history of another invasive malignancy within 3 years before the first dose of study drug that cannot be watched and requires treatment, or any evidence of residual disease from a previously diagnosed malignancy that cannot be watched and requires treatment. Adjuvant hormonal therapy for breast cancer is allowed.
* Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of enfortumab vedotin. Routine antimicrobial prophylaxis is permitted.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with enfortumab vedotin.
* History of idiopathic pulmonary fibrosis; organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Prior allogeneic stem cell or solid organ transplant.
* Other underlying medical condition that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study.
* Patients with active tuberculosis.
* Pregnant or breast feeding

EV/Pembrolizumab exploratory arm only:

* Patients who received prior immunotherapy for metastatic urothelial carcinoma (mUC) or for an alternative malignancy are eligible unless they developed an immune related adverse event while on therapy requiring cessation of therapy or use of disease modifying agents, corticosteroids, or immunosuppressive drugs.
* History of autoimmune diseases. Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

  * Patients with vitiligo or residual autoimmune hypothyroidism on stable doses of hormone replacement are permitted to enroll.
  * Patients with type 1 diabetes mellitus (T1DM) on a stable dose of insulin are permitted to enroll.
  * Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* On high dose steroids at the time of study enrollment, defined as >20mg prednisone (or bioequivalent), including steroids used for management of intracranial lesions. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Duration of clinical benefit | 8 months
  Duration of Clinical Benefit (DoCB) in patients undergoing EV schedule de-escalation in the EV monotherapy cohort. DoCB is defined as time from initiating treatment to disease progression or death in patients who achieve complete response, partial response, or stable disease (per RECIST v1.1)

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) in patients undergoing EV schedule de-escalation in the EV monotherapy cohort
Time to next treatment | 5 years
  Time to Next Treatment in patients undergoing EV schedule de-escalation in the EV monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Ghatalia, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No